CLINICAL TRIAL: NCT05538156
Title: Internal Limiting Membrane Peeling in Macula-off Retinal Detachment With Grade B Proliferative Vitreoretinopathy
Brief Title: Internal Limiting Membrane Peeling in Retinal Detachment Surgery
Acronym: IMPURITY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A00665-38
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-07

CONDITIONS: Retinal Detachment; Proliferative Vitreoretinopathy
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): The internal limiting membrane is not removed
  Interventions: Procedure: Control group
- Intervention group (Other): The internal limiting membrane of the posterior pole is removed
  Interventions: Procedure: Intervention group

INTERVENTIONS:
Procedure: Control group — Vitrectomy and gas tamponade without internal limiting membrane peeling
  Arms: Control group
Procedure: Intervention group — Vitrectomy, internal limiting membrane peeling and gas tamponade
  Arms: Intervention group

SUMMARY:
Despite advances in surgical techniques over the recent decades, proliferative vitreoretinopathy (PVR) remains the main obstacle to successful rhegmatogenous retinal detachment (RRD) repair, accounting for nearly 75% of all primary surgical failures. It is characterized by the growth and contraction of cellular membranes within the vitreous cavity and on both surfaces of the detached retina as well as intraretinal fibrosis.

The Retina Society classification, modified in 1991 and currently the most widely used, divided PVR into three grades. Grade A is limited to the presence of vitreous haze and pigment clumps. Grade B includes rolled or irregular edges of tear and/or inner retinal surface wrinkling with possible retinal stiffness and vessel tortuosity. Grade C is defined as the presence of full-thickness fixed retinal folds and is further subdivided based on the number of hours involved and the location.

Recently, Foveau et al., in a retrospective comparative case series, have demonstrated that performing internal limiting membrane (ILM) peeling during RRD surgery may increase the anatomical success rate for this indication.

The aim of this multi-center, prospective, randomized controlled clinical trial study is to evaluate the effectiveness of ILM peeling on surgical outcomes in patients with primary macula-off RRD complicated by grade B PVR.

DETAILED DESCRIPTION:
Despite advances in surgical techniques over the recent decades, proliferative vitreoretinopathy (PVR) remains the main obstacle to successful rhegmatogenous retinal detachment (RRD) repair, accounting for nearly 75% of all primary surgical failures. It is characterized by the growth and contraction of cellular membranes within the vitreous cavity and on both surfaces of the detached retina as well as intraretinal fibrosis.

The Retina Society classification, modified in 1991 and currently the most widely used, divided PVR into three grades. Grade A is limited to the presence of vitreous haze and pigment clumps. Grade B includes rolled or irregular edges of tear and/or inner retinal surface wrinkling with possible retinal stiffness and vessel tortuosity. Grade C is defined as the presence of full-thickness fixed retinal folds and is further subdivided based on the number of hours involved and the location.

Grade B PVR is thought to represent an immature form of PVR with a definite potential for progression to further stages of PVR. Specific treatment for moderate PVR seems to be essential to halt the disease process and to reduce the risk of postoperative re-detachment. However, there is currently no consensus regarding the management of grade PVR. In macula-off RRD, vitrectomy with gas tamponade is often used as a primary option, with a retinal reattachment rate of 60%.

Recently, Foveau et al., in a retrospective comparative case series, have demonstrated that performing internal limiting membrane (ILM) peeling during RRD surgery may increase the anatomical success rate for this indication.

The aim of this multi-center, prospective, randomized controlled clinical trial study is to evaluate the effectiveness of ILM peeling on surgical outcomes in patients with primary macula-off RRD complicated by grade B PVR.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* With macula-off retinal detachment complicated by grade B proliferative vitreoretinopathy

Exclusion Criteria:

* Underage patients
* History of retinal detachment
* History of intraocular surgery (except for cataract surgery)
* Traumatic retinal detachment
* Macular hole-associated retinal detachment
* Concurrent macular disease (diabetic maculopathy, age-related macular degeneration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary anatomical success rate | 12 months after surgery
  Primary retinal reattachment rate

SECONDARY OUTCOMES:
Functional outcomes #1 | 12 months after surgery
  Visual acuity (Logarithm of the Minimum Angle of Resolution)
Functional outcomes #2 | 12 months after surgery
  Degree of metamorphopsia (M-CHARTS)
Anatomical outcomes #1 | 12 months after surgery
  Integrity of the photoreceptor layer on Spectral Domain Optical Coherence Tomography
Anatomical outcomes #2 | 12 months after surgery
  Incidence of epiretinal membrane
Anatomical outcomes #3 | 12 months after surgery
  Incidence of cystoid macular edema
Anatomical outcomes #4 | 12 months after surgery
  Incidence of DONFL appearance
Functional outcomes #3 | 12 months after surgery
  Retinal sensitivity on microperimetry testing

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste CONART, Prof, Principal Investigator — Brabois Hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borowicz D, Nowomiejska K, Nowakowska D, Brzozowska A, Toro MD, Avitabile T, Junemann AG, Rejdak R. Functional and morphological results of treatment of macula-on and macula-off rhegmatogenous retinal detachment with pars plana vitrectomy and sulfur hexafluoride gas tamponade. BMC Ophthalmol. 2019 May 24;19(1):118. doi: 10.1186/s12886-019-1120-3. PMID 31126280
- [Result] Charteris DG. Proliferative vitreoretinopathy: pathobiology, surgical management, and adjunctive treatment. Br J Ophthalmol. 1995 Oct;79(10):953-60. doi: 10.1136/bjo.79.10.953. No abstract available. PMID 7488586
- [Result] Eissa MGAM, Abdelhakim MASE, Macky TA, Khafagy MM, Mortada HA. Functional and structural outcomes of ILM peeling in uncomplicated macula-off RRD using microperimetry & en-face OCT. Graefes Arch Clin Exp Ophthalmol. 2018 Feb;256(2):249-257. doi: 10.1007/s00417-017-3875-7. Epub 2018 Jan 3. PMID 29299741
- [Result] Fallico M, Russo A, Longo A, Pulvirenti A, Avitabile T, Bonfiglio V, Castellino N, Cennamo G, Reibaldi M. Internal limiting membrane peeling versus no peeling during primary vitrectomy for rhegmatogenous retinal detachment: A systematic review and meta-analysis. PLoS One. 2018 Jul 19;13(7):e0201010. doi: 10.1371/journal.pone.0201010. eCollection 2018. PMID 30024983
- [Result] Foveau P, Leroy B, Berrod JP, Conart JB. Internal Limiting Membrane Peeling in Macula-off Retinal Detachment Complicated by Grade B Proliferative Vitreoretinopathy. Am J Ophthalmol. 2018 Jul;191:1-6. doi: 10.1016/j.ajo.2018.03.037. Epub 2018 Apr 3. PMID 29621507
- [Result] Steel DH, Joussen AM, Wong D. ILM peeling in rhegmatogenous retinal detachment; does it improve the outcome? Graefes Arch Clin Exp Ophthalmol. 2018 Feb;256(2):247-248. doi: 10.1007/s00417-017-3876-6. Epub 2017 Dec 27. No abstract available. PMID 29282562